CLINICAL TRIAL: NCT03365921
Title: An Randomized, Double-blinded Trial of Recombinant Hepatitis E Vaccine (Escherichia Coli) Hecolin® to Evaluate Lot-to-lot Consistency
Brief Title: A Phase Ⅳ Clinical Trial of the Recombinant Hepatitis E Vaccine (Escherichia Coli)(the Lot Consistency Trial)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xiamen Innovax Biotech Co., Ltd (Industry)
Collaborators: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRO-HE-010
Record Dates: First submitted 2017-12-01; First posted 2017-12-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Hepatitis E
MeSH Terms: conditions — Hepatitis E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hepatitis E vaccine lot 1 (Experimental)
  Interventions: Biological: Participants would receive 3 doses of Recombinant Hepatitis E Vaccine (Escherichia Coli) intramuscularly at 0, 1, 6 month.
- Hepatitis E vaccine lot 2 (Experimental)
  Interventions: Biological: Participants would receive 3 doses of Recombinant Hepatitis E Vaccine (Escherichia Coli) intramuscularly at 0, 1, 6 month.
- Hepatitis E vaccine lot 3 (Experimental)
  Interventions: Biological: Participants would receive 3 doses of Recombinant Hepatitis E Vaccine (Escherichia Coli) intramuscularly at 0, 1, 6 month.

INTERVENTIONS:
Biological: Participants would receive 3 doses of Recombinant Hepatitis E Vaccine (Escherichia Coli) intramuscularly at 0, 1, 6 month. — Participants would receive 3 doses of Recombinant Hepatitis E Vaccine (Escherichia Coli) intramuscularly at 0, 1, 6 month.

SUMMARY:
This study is to evaluate lot-lot consistency of Recombinant Hepatitis E Vaccine (Escherichia Coli) Hecolin®.

DETAILED DESCRIPTION:
This study is a mono-center, randomization, double-blind clinical trial in healthy subjects between 18 to 50. Under the premise of full informed consent, 360 subjects that meet the requirement of clinical trial in the age of 18-50 will be divided into 3 groups and injected 3 consecutive batches of Hecolin® separately. The main outcome measures are the immunogenicity evaluation and safety surveillance after inoculation according to prescribed immunization procedure.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged over 18 years old to 50 years old on the day of enrollment 2. Axillary temperature is below than 37.0 ℃. 3.Negative serological markers for hepatitis E 4. Judged as healthy and eligible for vaccination by the investigators through a selfreported medical history and some physical examinations.

  5. Able to understand this study information and willing to comply with all study requirements.

  6. Willing to participate in this study and sign informed consent form.

Exclusion Criteria:

1. Pregnancy,breast-feeding or plan to be pregnant in 7 months;
2. Administration of Hepatitis E Vaccine before the study;
3. Participate in any other clinical trial during the study period;
4. Use of any investigational product or non-registered product (drug or vaccine)within 30 days preceding the first dose of the study vaccine or plan to use during the study period;
5. Received immunosuppressed, immunoregulation therapy or corticosteroid systemic therapy for more than 14 days in the 6 months before entry, except local treatment;
6. Administration of any immunoglobulin or blood products within 3 months preceding the first dose of the study vaccine,or plan to use during the study period;
7. Administration of any inactivated vaccines within 14 days preceding the first dose of the study or attenuated live vaccines within 21 days preceding the first dose of the study;
8. Had a fever (axillary temperature over 38°C) within 3 days or acute illness, or use systemic antibiotics or antiviral treatment within 5 days before vaccination;
9. Immunodeficiency (such as HIV carriers), primary disease of important organs, malignant tumor, or any immune disease (such as systemic lupus erythematosus, arthritis pauperum, splenectomy or functional asplenia or other disease which might affect immune response), liver and kidney disease and other chronic disease history;
10. History of allergic disease or history of serious adverse events occurring after vaccination, i.e., allergy,urticaria, dyspnea, angioneurotic edema or abdominal pain. Allergic history to any component of this vaccine.

12. Asthma that needed emergency treatment, hospitalization, oral or intravenous corticosteroid to keep stable in the past two years; 12. Combining another severe internal medicine disease(such as cardiopathy,diabetes and hyperthyroidism) 13. Anormal coagulation function or coagulopathy diagnosed by doctor; 14. Epilepsy(not including alcohol epilepsy within 3 years prior to abstinence and simple epilepsy that do without curing within 3 years prior to the study ) 15. Anomal psychology or mind affecting the individual's ability to obey the study requirement; 16. Other medical, psychological, social or occupational factors that, according to the investigators' judgment,might affect the individual's ability to obey the protocol or sign the informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 360 (Actual)
Dates: Start 2018-10-27 (Actual); Primary Completion 2019-06-16 (Actual); Study Completion 2019-06-16 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate and GMC of anti-HEV IgG at Month 7. | 7 months
  Measure anti-HEV IgG in serum samples at 7 month to evaluate the immunogenicity of the Hepatitis E vaccine.

SECONDARY OUTCOMES:
Adverse reactions/events of all subjects | up to 7 months
  Measure solicited local adverse reactions within 7 days after each vaccination; Measure solicited systematic adverse reactions within 7 days after each vaccination; Measure unsolicited adverse reactions within 30 days after vaccination; Measure serious adverse events occurred throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Yuemei Hu, Principal Investigator — Jiangsu Provincial Center for Disease Prevention and Control
Locations (1):
- Dongtai City Center for Disease Control and Prevention, Dongtai, Jiangsu, China